CLINICAL TRIAL: NCT05869968
Title: Biomarkers of Immune Dysfunction and Vaccine Responsiveness in People With Chronic Traumatic Spinal Cord Injury
Brief Title: SCIVAX: Biomarkers of Immune Dysfunction and Vaccine Responsiveness in Chronic SCI
Acronym: SCIVAX
Status: Recruiting | Type: Observational
Sponsor: Northwell Health (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); New York State Department of Health (Other Government)
Responsible Party: Principal Investigator, Ona Bloom, Professor, Northwell Health
Other Study IDs: 22-0787-FIMR
Record Dates: First submitted 2023-05-10; First posted 2023-05-23 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Spinal Cord Injuries; Traumatic Spinal Cord Injury; Healthy Controls; Flu Vaccine; COVID-19 Vaccine
Keywords: Chronic Spinal Cord Injury; Flu Vaccination; COVID-19 Vaccination; Immune Responsiveness
MeSH Terms: conditions — Spinal Cord Injuries; Influenza, Human

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and a self-collected nasal swab will be collected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Individuals with Chronic Spinal Cord Injury who receive either Flu or COVID-19 vaccine: 18-89 years old with traumatic SCI, AIS grade A-D, Neurological injury level of C1-T10 who are choosing to receive a vaccine against the flu or COVID-19 and demonstrate capacity to provide informed consent.
- Uninjured Controls who receive the Flu vaccine or COVID-19 vaccine: 18-89 years old without traumatic Spinal Cord Injury (SCI) who are choosing to receive a vaccine against either the Flu or COVID-19 and demonstrate the capacity to provide informed consent.

SUMMARY:
The purpose of this observational research study is to better understand immune responses to vaccines against viruses (influenza or SARS-CoV2). The goal is to determine any differences in immune responses to vaccines in uninjured people and in people living with spinal cord injuries, who are typically at increased risk of infections.

DETAILED DESCRIPTION:
The purpose of this research study is to measure a person's immune response to a vaccine by measuring types of circulating white blood cells (WBC) and the substances they produce in blood, including antibodies, proteins, and ribonucleic acids (the body's genetic blueprint for making proteins).

The research will study two populations: uninjured people and people living with spinal cord injury (SCI), who are often at increased risk of infections. We will measure and observe over time any differences in immune responses to vaccines between those groups or among people with SCI according to their injury severity or level.

The overall goal of this study is to increase knowledge of immune responses to vaccination against influenza virus that causes the flu, and to the SARS-CoV-2 virus that causes COVID-19. There is currently a lack of information about what influences individual responses to vaccines and why people with SCI are at typically at increased risk of infection. Results from this study may teach us how to improve vaccination strategies and other ways to fight infections in uninjured people and in people with SCI

ELIGIBILITY:
Inclusion Criteria

SCI Participant Inclusion Criteria: To be eligible for prospective enrollment, participants are required to meet the following inclusion criteria:

* 18-89 years old with traumatic SCI
* initial traumatic SCI >/=1 year from enrollment (DOD funded study)
* initial traumatic SCI <1 year from enrollment (non-DOD funded pilot study)
* American Spinal Injury Association (ASIA) classification grade A-D
* Neurological Injury Level C1-T10
* Demonstrate capacity to provide informed consent using the "teach back" method to verify understanding and appreciation of study objectives and procedures.

Exclusion Criteria

To be eligible for prospective enrollment, SCI participants are required to not meet the following exclusion criteria:

* Stage III-IV pressure ulcers
* Cancer, chemotherapy, neutropenia
* Pregnancy or lactation
* No known SCI
* Autoimmune disease
* Pre-existing neurological disease
* History of dementia
* Any other condition that would compromise their ability to provide informed consent
* Any other condition that a study physician feels would preclude participation or be contraindicated

Uninjured Control Group:

Inclusion Criteria

Uninjured Control Participant Inclusion Criteria: To be eligible for prospective enrollment, participants are required to meet the following inclusion criteria:

* 18-89 years old without traumatic SCI
* Demonstrate capacity to provide informed consent using the "teach back" method to verify understanding and appreciation of study objectives and procedures.

Exclusion Criteria

To be eligible for prospective enrollment, uninjured control participants are required to not meet the following exclusion criteria:

* Cancer, chemotherapy, neutropenia
* Pregnancy or lactation
* Autoimmune disease
* Pre-existing neurological disease
* History of dementia
* Any other condition that would compromise their ability to provide informed consent
* Any other condition that a study physician feels would preclude participation or be contraindicated

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be adults (ages 18-89 years old) with SCI or who are uninjured controls who are electing to receiving flu or COVID-19 vaccines to promote their health.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2023-03-31 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
mRNA transcript levels for genes expressed according to white blood cell type after flu vaccination | 0-28 days after flu vaccination
  Serum samples will be used to determine if gene expression levels made by specific types of white blood cells are different between participant groups and within the SCI group by injury level and severity.
Anti-flu antibody titers in response to vaccination | 0-28 days after flu vaccination
  Serum samples will be used to determine antibody titers for anti-flu antibodies at baseline and after vaccination. These samples will be obtained to determine if vaccine responses are different between participant groups and within the SCI group by injury level and severity

SECONDARY OUTCOMES:
mRNA transcript levels for genes expressed according to white blood cell type after COVID-19 vaccination | 0-28 days after COVID-19 vaccination
  Serum samples will be used to determine if gene expression levels made by specific types of white blood cells are different between participant groups and within the SCI group by injury level and severity.
Anti-COVID-19 antibody titers in response to vaccination | 0-28 days after COVID-19 vaccination
  Serum samples will be used to determine antibody titers for anti-COVID-19 antibodies at baseline and after vaccination. These samples will be obtained to determine if vaccine responses are different between participant groups and within the SCI group by injury level and severity
Systemic inflammatory cytokine levels in response to vaccination | 0-28 days after vaccination
  Serum samples will be used to determine systemic inflammatory cytokine levels at baseline and after flu or COVID-19 vaccination. These samples will be obtained to determine if cytokine levels are different between participant groups and within the SCI group by injury level and severity

CONTACTS AND LOCATIONS:
Overall Officials: Ona Bloom, PhD, Principal Investigator — Feinstein Institute for Medical Research; Northwell Health
Locations (1):
- Northwell Health, Manhasset, New York, United States